CLINICAL TRIAL: NCT05510713
Title: Preliminary Study on the Effect of Blood Purification Therapy With Dual-cannula in Jugular-femoral Venous
Brief Title: Blood Purification Therapy With Dual-cannula in Jugular-femoral Venous
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: jv-fv-RRT
Record Dates: First submitted 2022-08-18; First posted 2022-08-22 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Blood Purification; Dual-cannula; Vena Cava Disconnection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the treatment-as-usual group (No Intervention): we used the single-cannula in femoral venous blood purification therapy in the following patients with vena cava disconnection or severe obstruction
- intervention group (Experimental): we used the dual-cannula in jugular-femoral venous blood purification therapy in the following patients with vena cava disconnection or severe obstruction
  Interventions: Device: Hemodialysis Catheter

INTERVENTIONS:
Device: Hemodialysis Catheter — We add a dialysis catheter to the patient, i.e., replace single-cannula in femoral venous with dual-cannula in jugular-femoral venous
  Arms: intervention group

SUMMARY:
Acute kidney failure (AKI) is one of the most important causes of morbidity and mortality for critical ill patients. The use of blood purification treatment such as renal replacement therapy (CRRT) and plasma exchange has gradually developed into an effective treatment. However, the efficiency of blood purification may be affected by the recirculation of dual-lumen venous catheter for some special patients including patients with vena cava reflux disorder from massive occupations or ascites. For extreme cases like patients with vena cava disconnection or severe obstruction, the traditional blood purification treatment cannot work effectively. Thus, we used the dual-cannula in jugular-femoral venous blood purification therapy in the following two patients and found that it can improve the perfusion of systemic circulation and the prognosis of patients

ELIGIBILITY:
Inclusion Criteria:

* 1. patients requiring haemodilution therapy for various reasons (acute renal failure, acute liver failure, etc.)
* 2. presence of superior vena cava and/or inferior vena cava reflux disorders
* 3. age greater than 18 years

Exclusion Criteria:

* 1. Inability to establish suitable vascular access
* 2. Pregnant women
* 3. Not agreeing to active life support treatment
* 4. Severe active bleeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
vasoactive drugs | 144 hours after dual-cannula in jugular-femoral venous
  doses of vasoactive drugs
ICU mortality | 28-day ICU mortality
  Measurement of ICU mortality

SECONDARY OUTCOMES:
Cytokine | 24hous after dual-cannula in jugular-femoral venous
  Checking cytokine levels by laboratory

CONTACTS AND LOCATIONS:
Overall Officials: Minjie Ju, PHD, Study Director — Shanghai Zhongshan Hospital

IPD SHARING:
Plan to Share IPD: No